CLINICAL TRIAL: NCT00424866
Title: A Phase 1, Open Label, Dose Response, Pilot Study to Evaluate the Safety and Tolerability of Human Fibroblast Growth Factor-1 (FGF-1) in Peripheral Arterial Disease Patients With Intermittent Claudication
Brief Title: FGF-1 for Intramuscular Injection for the Treatment of Peripheral Arterial Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CardioVascular BioTherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVBT-2006-PAD-01
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Arterial Disease; Stenosis; Intermittent Claudication
Keywords: Peripheral Arterial Disease; Ischemia; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Constriction, Pathologic; Intermittent Claudication; Ischemia | interventions — Fibroblast Growth Factor 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The dosing groups correspond to total doses of 0 µg/kg of FGF-1.
  Interventions: Drug: Placebo
- Human FGF-1 (Active Comparator): The dosing groups correspond to total doses of either 3, 10 or 30 µg/kg of FGF-1.
  Interventions: Drug: FGF-1

INTERVENTIONS:
Drug: FGF-1 — Doses of FGF-1: 3 ug/kg; 10 ug/kg; 30 ug/kg
  Low dose: 3.0 μg/kg Mid dose: 10 μg/kg High dose: 30 µg/kg
  Other Names: Acidic FGF
  Arms: Human FGF-1
Drug: Placebo — Vehicle: 0 µg/kg
  Arms: Placebo

SUMMARY:
FGF-1 for the treatment of patients with peripheral arterial disease with intermittent claudication.

DETAILED DESCRIPTION:
FGF-1 administered by intramuscular injection for the treatment of peripheral arterial disease with intermittent claudication. Eligible patients are allocated to one of three treatment arms. Patients within each dosing group will be randomized between study drug and vehicle control. Safety, pharmacokinetics, and cardiovascular improvement will be evaluated at day 1 and weeks 1, 4 and 12 post dosing.

ELIGIBILITY:
Inclusion Criteria

1. Subjects considered eligible to enter the study must sign an informed consent form prior to the initiation of any study procedures. In the event that the subject must be withdrawn and is re-screened for study participation at a later date, a new informed consent form must be signed. Subjects must be competent to give written informed consent.
2. Age must be ≥50 and ≤75 years of age with a life expectancy of > 1 year and leg survival > 6 months. Patients >75 and ≤80 years of age will be considered if they show no signs of cognitive or muscle function decline and are fully able to comply with the protocol.
3. Patients must have experienced intermittent claudication for at least 6 months and have been stable for the past 3 months.
4. Patients must have peripheral arterial disease, as confirmed by a resting ABI ≥0.40 and <0.90 based on at least one leg as measured using both the dorsal pedis and posterior tibial arteries.
5. Stenosis of >70% up to total occlusion must be present in the popliteal artery and/or in the tibial peroneal trunk or at least 2 tibial arteries above the ankle without inflow limitation of the popliteal artery. Adequate popliteal inflow is defined as continuous flow from the abdominal aorta, iliac, common femoral and superficial femoral with any stenosis < 50% as determined either by intra-arterial DSA, CTA or Gd CE-MRA.
6. The screening Gardner treadmill test peak walking times (PWT) must be >1 minute and < 12 minutes and limited by pain in one or both calves.
7. Preexisting medication regime must be stable for 6 weeks preceding dosing.

Exclusion Criteria

1. Evidence of critical leg ischemia, i.e. ischemic rest pain or ischemic ulceration
2. Treadmill walking limited by conditions other than intermittent claudication including arthritis, angina and dyspnea
3. Lower limb amputation of, or in, either leg including toes
4. Evidence of limb ischemia from immunologic or inflammatory disorders
5. Leg surgery or revascularization within past 6 months or peripheral angioplasty within past 3 months or anticipated during study
6. Participation in any investigational device or drug trial within the past 6 months
7. Myocardial infarction, unstable angina, stroke or ischemic attack within past 6 months
8. New York Heart Association (NYHA) class II, III or IV heart failure, restrictive or hypertrophic cardiomyopathy or severe valvular disease
9. QTc elongation greater than 450 ms in males or 460 ms in females
10. PT (INR), PTT, urinalysis, thyroid function (T3, T4, TSH) outside normal limits
11. Hemorrhage or thrombotic events (e.g. deep vein thrombosis) within past 6 months
12. Thrombocytopenia (<100,000/µl), history of heparin-induced thrombocytopenia
13. Major surgery with the past 6 months
14. Positive proliferative retinopathy exam
15. Present of any type of cancer or history of cancer except past (but not present) basal cell dermal carcinoma not on either leg
16. Inflammatory or progressive fibrotic or myelofibrotic disorders
17. Patients experiencing bacterial or viral infection (e.g. hepatitis or HIV) or who may otherwise be febrile
18. Hemoglobin A1c(HgbA1c) of >8%
19. Type I diabetes
20. Total fasting cholesterol >200
21. Uncontrolled hypertension (≥160 systolic or ≥100 diastolic pressure) or hypotension (<90 systolic or <60 diastolic pressure)
22. Disease or drug (e.g. systemic corticosteroid) immuno-compromised
23. Hepatic dysfunction as defined either by AST or ALT > 2.0 times the upper limit of normal
24. Serum creatinine of ≥ 2.5 mg/dl
25. Proteinuria (urine protein/creatinine ratio > 3)
26. Antiproliferative drugs (e.g. thalidomide, hydroxyurea)
27. Radiation therapy
28. Implanted devices not compatible with strong magnetic fields
29. Life expectance of less than 1 year
30. Females who are premenopausal and not sterilized or using adequate birth control or are either pregnant, intend to become pregnant or are nursing

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of i.m. injected Cardio Vascu Grow TM, a recombinant Human Fibroblast Growth Factor-1 (FGF-1-141) | From enrollment through study completion, an average of 12 weeks
  Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs)
Change from baseline in safety laboratory measurements at 12 weeks | From enrollment through study completion, an average of 12 weeks
  Safety laboratory evaluations on hematology, serum chemistry, and urinalysis

SECONDARY OUTCOMES:
Plasma FGF-1 (1-141) pharmacokinetic measurements at pre-dose, 5, 15, and 30 minutes and at 1, 2, 4, 6, 10, and 24 hours | From enrollment through study completion, an average of 12 weeks
  Pharmacokinetic plasma concentrations of FGF-1 (1-141)

CONTACTS AND LOCATIONS:
Locations (1):
- CVBT Info, Dallas, Texas, United States